CLINICAL TRIAL: NCT01433250
Title: An Open Label Extension Study to Evaluate the Safety, Tolerability and Efficacy of AIN457 in Patients With Relapsing-remitting Multiple Sclerosis
Brief Title: A Study to Evaluate the Safety, Tolerability and Efficacy of AIN457 in Patients With Relapsing-remitting Multiple Sclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAIN457B2201E1; 2011-001629-25 (EudraCT Number)
Record Dates: First submitted 2011-08-26; First posted 2011-09-13 (Estimated); Results first posted 2016-03-14 (Estimated); Last update posted 2016-03-14 (Estimated); Status verified 2016-02

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis,; demyelinating autoimmune diseases,; interleukin-17,; monoclonal human antibody
MeSH Terms: conditions — Multiple Sclerosis | interventions — secukinumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- AIN 457 Core (Experimental): (10mg/kg i.v.). AIN 457 core study /AIN 457 Extension
  Interventions: Drug: AIN457
- AIN457 Placebo Core (Experimental): (10mg/kg i.v.). AIN 457 placebo core study /AIN 457 Extension
  Interventions: Drug: AIN457

INTERVENTIONS:
Drug: AIN457 — (10mg/kg i.v.).
  Other Names: AIN457 core/ AIN extension
  Arms: AIN 457 Core
Drug: AIN457 — (10mg/kg i.v.).
  Other Names: AIN Placebo / AIN Extension
  Arms: AIN457 Placebo Core

SUMMARY:
The study will assess the long-term safety and tolerability of AIN457 in patients with relapsing-remitting multiple sclerosis (RRMS). In addition the long-term pattern of maintenance of efficacy and health related quality of life will be explored.

ELIGIBILITY:
Inclusion Criteria:

1. Was exposed to AIN457 or placebo in study CAIN457B2201 and completed the CAIN457B2201 study, up to at and including Visit 10 (week 24).

Exclusion Criteria:

1. Have been treated with:

   * immunosuppressive medications such as azathioprine or methotrexate within 1 month prior to enrollment, if lymphocyte count normal.
   * immunoglobulins and/or monoclonal antibodies (with the exception of AIN457) within 2 month prior to enrollment, or if the immunosuppressive effects are likely to persist at enrollment (such as presence of B cell depletion after rituximab treatment).
2. Have received total lymphoid irradiation, bone marrow transplantation, alemtuzumab, cladribine, cyclophosphamide, mitoxantrone or other immunosuppressive treatments with long-lasting (over 6 months) or permanent effects.
3. Have received any live or live attenuated vaccines (including live vaccines for varicella-zoster virus or measles) within 2 months prior to enrollment.
4. A diagnosis of chronic disease of the immune system other than MS, or of an immunodeficiency syndrome.
5. Current severe depression.
6. Pregnant or nursing (lactating) women.
7. Malignancy diagnosed since enrollment in the core study (except for successfully-treated basal or squamous cell carcinoma of skin).
8. A new diagnosis of diabetes
9. Positive testing for tuberculosis (QuantiFeron or chest X-ray).
10. Subjects with clinically significant cardiac abnormalities
11. Unable or unwilling to undergo multiple venipunctures
12. Unable to undergo MRI scans due to newly acquired claustrophobia or metallic implants incompatible with MRI.

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2012-02; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (13):
- Czechia (5):
  - Novartis Investigative Site, Hradec Králové, Czech Republic
  - Novartis Investigative Site, Ostrava
  - Novartis Investigative Site, Ostrava-Moravska Ostrava
  - Novartis Investigative Site, Prague
  - Novartis Investigative Site, Teplice
- Russia (4):
  - Novartis Investigative Site, Kazan'
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Nizhny Novgorod
  - Novartis Investigative Site, Smolensk
- Ukraine (4):
  - Novartis Investigative Site, Kharkiv
  - Novartis Investigative Site, Kiev
  - Novartis Investigative Site, Odesa
  - Novartis Investigative Site, Vinnitsya

RESULTS

PARTICIPANT FLOW:
Groups:
- AIN457 Core / AIN457 Extension: AIN in core study , continued AIN in extension study ( 10 mg/Kg iv every four weeks)
- AIN Placebo/ AIN457 Extension: Placebo in core study and AIN in extension study
  (10 mg/kg iv every four weeks)
Period: Overall Study
Arm/Group | AIN457 Core / AIN457 Extension | AIN Placebo/ AIN457 Extension
Started | 22 | 17
Completed | 19 | 14
Not Completed | 3 | 3
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- AIN457/ AIN457: AIN in core study , continued AIN in extension study
- Placebo/AIN457: Placebo for core study and AIN in extension study
- Total: Total of all reporting groups
Arm/Group | AIN457/ AIN457 | Placebo/AIN457 | Total
Number analyzed (Participants) | 22 | 17 | 39
Age, Continuous [Mean (Standard Deviation); unit: Years] | 36.1 (10) | 34.2 (8.71) | 35.3 (9.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 12 | 24
  Male | 10 | 5 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 20 | 16 | 36
  Unknown or Not Reported | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Measure: Number of Subjects With Adverse Events, Number of Abnormalities in Safety Assessments
Description: Safety outcomes will be described in Adverse events section as there was not an efficacy primary outcome
Time Frame: 97 weeks
Measure: Number; unit: participants
Groups:
- AIN/AIN: AIN core 24 weeks/AIN extension 1 year
- PBO/AIN: placebo first 24 weeks/ AIN extension for 52 weeks
Arm/Group | AIN/AIN | PBO/AIN
Number analyzed (Participants) | 22 | 17
participants | 12 | 8

2. Secondary Outcome: Distribution of Patients With Relapses to End of Study (EOS) (All Subjects)
Description: Description: number of relapses based on neurological assessments and EDSS
Time Frame: week 97
Measure: Number; unit: Participants
Arm/Group | AIN/AIN | PBO/AIN
Number analyzed (Participants) | 22 | 17
Participants | 9 | 5

3. Secondary Outcome: Number Lesions Measured in the Brain by Magnetic Resonance Imaging. T1 Weighted MRI
Description: Measures of absolute number of gadolinium [Gd]-enhancing lesions on T1-weighted scans
Time Frame: weeks 13,25,37,53,73 and 97
Measure: Mean (Full Range); unit: lesions
Arm/Group | AIN/AIN | PBO/AIN
Number analyzed (Participants) | 22 | 17
lesions
  week 13 T1 (n=22, 16) | 0.8 [0.0 to 4.0] | 2.0 [0.0 to 15]
  week 25 T1 (n=22, 16) | 0.6 [0.0 to 5.0] | 1.9 [0 to 20]
  week 37 T1 (n=22, 15) | 1.0 [0.0 to 5.0] | 0.8 [0.0 to 4.0]
  week 53 T1 (n=14, 6) | 0.3 [0.0 to 3.0] | 0.3 [0.0 to 1.0]
  wk 73 T1 (n=11,9) | 0.6 [0.0 to 3.0] | 0.2 [0.0 to 1.0]
  EOT (n=15,13) | 0.7 [0.0 to 5.0] | 0.5 [0.0 to 3.0]

4. Secondary Outcome: Number Lesions Measured in the Brain by Magnetic Resonance Imaging. T2 Weighted MRI
Description: Measures of absolute number of gadolinium [Gd]-enhancing lesions on T2-weighted lesions
Time Frame: weeks 13,25,37,53,73 and 97
Measure: Mean (Full Range); unit: lesions
Arm/Group | AIN/AIN | PBO/AIN
Number analyzed (Participants) | 22 | 17
lesions
  week 13 T2 (n=22, 16) | 1.3 [0.0 to 7.0] | 2.2 [0.0 to 12.0]
  week 25 T2 (n=22, 16) | 0.8 [0.0 to 6.0] | 2.4 [0 to 21]
  week 37 T2 (n=22, 15) | 1.3 [0.0 to 5.0] | 1.3 [0.0 to 6.0]
  week 53 T2 (n=14, 6) | 0.4 [0.0 to 4.0] | 0.7 [0.0 to 3.0]
  wk 73 T2 (n=11,9) | 1.3 [0.0 to 5] | 0.9 [0.0 to 5.0]
  EOT T2 (n=15,13) | 1.1 [0.0 to 4.0] | .07 [0.0 to 3.0]

5. Secondary Outcome: Change in Brain Volume at End of Study.
Description: Change in volume from start to end of study
Time Frame: week 97
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | AIN/AIN | PBO/AIN
Number analyzed (Participants) | 22 | 17
ml | -14.8968 (63.73027) | -30.4346 (31.21800)

6. Secondary Outcome: Measure of Disability: Expanded Disability Status Scale (EDSS).
Description: The EDSS is a scale for assessing neurological impairment in MS (Kurtzke 1983) including (1) a series of scores in each of eight functional systems, and (2) the EDSS steps (ranging from 0 (normal) to 10 (death due to MS). The functional systems are Visual, Brain Stem, Pyramidal, Cerebellar, Sensory, Bowel and Bladder, Cerebral and Other functions.
Time Frame: Baseline to week 97
Population: Not all patients may have been available at all time points for EDSS evaluation
Measure: Number; unit: participants
Arm/Group | AIN/AIN | PBO/AIN
Number analyzed (Participants) | 22 | 17
participants
  Baseline score 0 | 1 | 0
  Baseline score 1.0 | 0 | 2
  Baseline score 1.5 | 5 | 5
  Baseline score 2.0 | 5 | 2
  Baseline score 2.5 | 1 | 1
  Baseline score 3.0 | 2 | 4
  Baseline score 3.5 | 2 | 0
  Baseline score 4.0 | 1 | 1
  Baseline score 4.5 | 2 | 2
  Baseline score 5.0 | 1 | 0
  Baseline score 6.0 | 1 | 0
  WK25 score 0 | 2 | 0
  WK25 score 1 | 1 | 2
  WK25 score 1.5 | 4 | 5
  WK25 score 2.0 | 4 | 1
  WK25 score 2.5 | 2 | 1
  WK25 score 3.0 | 2 | 4
  WK25 score 4.0 | 1 | 1
  WK25 score 4.5 | 3 | 1
  WK25 score 5.0 | 1 | 0
  WK25 score 5.5 | 0 | 1
  WK25 score 6.0 | 1 | 0
  WK25 score 6.5 | 1 | 0
  Safety Week 53 score 0 | 1 | 0
  Safety Week 53 score 1.0 | 1 | 1
  Safety Week 53 score 1.5 | 3 | 3
  Safety Week 53 score 2.0 | 4 | 0
  Safety Week 53 score 3.0 | 1 | 1
  Safety Week 53 score 3.5 | 1 | 0
  Safety Week 53 score 4.0 | 0 | 1
  Safety Week 53 score 5.0 | 1 | 0
  Safety Week 53 score 5.5 | 2 | 0
  Safety Week 53 score 6.0 | 1 | 0
  WK73 score 0 | 1 | 1
  WK73 score 1.0 | 2 | 1
  WK73 score 1.5 | 1 | 5
  WK73 score 2.0 | 2 | 0
  WK73 score 3.0 | 0 | 1
  WK73 score 4.0 | 1 | 0
  WK73 score 5.5 | 1 | 0
  WK73 score 6.0 | 1 | 0
  End of treatment score 0 | 1 | 1
  End of treatment score1.0 | 2 | 1
  End of treatment score 1.5 | 2 | 5
  End of treatment score 2.0 | 2 | 1
  End of treatment score 2.5 | 2 | 1
  End of treatment score 3.0 | 0 | 3
  End of treatment score 3.5 | 1 | 0
  End of treatment score 4.0 | 2 | 0
  End of treatment score 4.5 | 0 | 1
  End of treatment score 5.5 | 0 | 1
  End of treatment score 6.0 | 1 | 0

ADVERSE EVENTS:
Groups:
- Placebo(Core)/AIN457(Extension): Placebo(core)/AIN457(extension)
- AIN457(Core)/AIN457(Extension): AIN457(core)/AIN457(extension)
Arm/Group | Placebo(Core)/AIN457(Extension) | AIN457(Core)/AIN457(Extension)
Serious Adverse Events (participants affected / at risk) | 0/17 | 2/22
Other Adverse Events (participants affected / at risk) | 8/17 | 7/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo(Core)/AIN457(Extension) (N=17) | AIN457(Core)/AIN457(Extension) (N=22)
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo(Core)/AIN457(Extension) (N=17) | AIN457(Core)/AIN457(Extension) (N=22)
Angina pectoris (Cardiac disorders) | 1 | 0
Cardiomyopathy (Cardiac disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Cystitis (Infections and infestations) | 1 | 0
Laryngitis (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 1
Pharyngitis (Infections and infestations) | 0 | 2
Respiratory tract infection viral (Infections and infestations) | 1 | 2
Rhinitis (Infections and infestations) | 1 | 0
C-reactive protein increased (Investigations) | 1 | 0
Overweight (Metabolism and nutrition disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Migraine (Nervous system disorders) | 1 | 0
Anxiety disorder (Psychiatric disorders) | 0 | 2
Uterine cervical erosion (Reproductive system and breast disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Hypertension (Vascular disorders) | 1 | 0
Varicose vein (Vascular disorders) | 0 | 2

LIMITATIONS AND CAVEATS:
Further development of secukinumab in MS is not being pursued and the extension study , CAIN457B2201E1, further enrollment stopped . Not completing enrollment of this study was not related to the safety or tolerability concerns observed in the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial